CLINICAL TRIAL: NCT07131683
Title: Human Umbilical Cord Mesenchymal Stem Cell-derived ExoSomes for Autoimmune Encephalitis: a Phase I/IIa Clinical Trial (MESAE)
Brief Title: hUC-MSC-Exo Therapy for Autoimmune Encephalitis
Acronym: MESAE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: ECHO Biotech (Unknown)
Responsible Party: Principal Investigator, cuilili, Principle investigator, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KS2025069; BRWEP2024W022010110 (Other Grant/Funding Number: Beijing Municipal Health Commission)
Record Dates: First submitted 2025-08-07; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Encephalitis
Keywords: mesenchymal stem cell; exosome; autoimmune encephalitis; safety; efficacy
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exosome group (Experimental)
  Interventions: Biological: Human umbilical cord mesenchymal stem cell derived exosomes
- Control group (Placebo Comparator)
  Interventions: Other: Placebo Control

INTERVENTIONS:
Biological: Human umbilical cord mesenchymal stem cell derived exosomes — Nasal spray of hUC-MSC-Exo (low dose: 2.5×10^10 particles, mid-dose: 5.0×10^10 particles, high-dose: 1.0×10^11 particles), once per day for 7 days, then once per week for 3 weeks
  Other Names: hUC-MSC-Exo
  Arms: Exosome group
Other: Placebo Control — Nasal spray of placebo control, once per day for 7 days, then once per week for 3 weeks
  Other Names: hUC-MSC-Exo mimics
  Arms: Control group

SUMMARY:
This is a phase I/IIa study to investigate the safety and preliminary efficacy of intranasal admnistration of human umbilical mesenchymal stem cell-derived exosome (hUC-MSC-Exo) for patients with autoimmune encephalitis.

DETAILED DESCRIPTION:
Dose Escalation Phase:

A multicenter, single-arm, open-label study will be conducted to evaluate the safety, tolerance, and dose exploration of multiple administrations of hUC-MSC-Exo for treating AE. Three dose cohorts (2.5×10¹⁰, 5.0×10¹⁰, and 1.0×10¹¹ particles) will be enrolled with 3-6 subjects each. Administration will be intranasal, once daily for 7 consecutive days, followed by once weekly for 3 consecutive weeks, resulting in a total treatment period of 4 weeks. After the last subject in each cohort completes the final dose and undergoes a 21-day safety assessment, a decision will be made regarding progression to the next higher dose cohort for further evaluation of safety and tolerance. The maximal tolerance dose (MTD) will be determined.

Case Expansion Phase:

A multicenter, randomized, double-blind, placebo-controlled study will enroll 20 subjects randomly assigned to either the experimental group (exosome group) or the control group (exosome mimetic group) in a 1:1 ratio. The dosage for the experimental group will be determined by the Data Safety Monitoring Board (DSMB) based on the safety and efficacy data obtained during the dose exploration phase.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years, both male and female are eligible;
2. Diagnosis of autoimmune encephalitis within 3 months of onset (meeting the 2016 Graus and Dalmau diagnostic criteria), with positive serum/cerebrospinal fluid anti-NMDAR antibodies or anti-LGI1 antibodies;
3. Modified Rankin Scale (mRS) score ≥ 2 at enrollment;
4. The subject or legally authorized representative is able to sign the informed consent form;
5. Subjects of childbearing potential must agree to practice strict contraception during the study period.

Exclusion Criteria:

1. Pre-morbid modified Rankin Scale (mRS) score ≥ 2;
2. Known allergy to any component of the investigational product or history of severe allergic reactions;
3. Presence of neurological or psychiatric disorders (e.g., cerebrovascular disease, Parkinson's disease, severe depression) deemed by the investigator to potentially impair trial participation or study assessments;
4. Current or history of any clinically significant systemic diseases judged by the investigator as unsuitable for inclusion, including but not limited to:

   * Severe cardiovascular diseases (e.g., congestive heart failure, severe arrhythmia, myocardial infarction)
   * Hepatic diseases (e.g., cirrhosis)
   * Renal diseases (e.g., requiring hemodialysis or peritoneal dialysis)
   * Hematological diseases (e.g., hemophilia with bleeding tendency)
   * Endocrine disorders (e.g., poorly controlled diabetes with blood glucose >16.8 mmol/L or <2.8 mmol/L, or with severe complications)
   * Immune system disorders (active or uncontrolled systemic autoimmune diseases, primary/secondary immunodeficiency)
   * Malignancies;
5. Anatomical nasal abnormalities, nasal mucosal damage, severe rhinitis, or other nasal conditions affecting drug administration;
6. Requiring nasogastric tube placement;
7. Organ function meeting any of the following criteria:

   1. Absolute neutrophil count (ANC) <1.5×10⁹/L, platelets (PLT) <100×10⁹/L, hemoglobin (Hb) <90 g/L
   2. Aspartate aminotransferase (AST) >2.5×ULN and/or alanine aminotransferase (ALT) >2.5×ULN, total bilirubin (TBIL) >1.5×ULN
   3. Creatinine >1.5×ULN
   4. Without anticoagulant/antiplatelet therapy: International normalized ratio (INR) >1.7 or activated partial thromboplastin time (APTT) >1.25×ULN With anticoagulant/antiplatelet therapy: INR >3.0 or APTT >1.5×ULN;
8. Positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with detectable HBV-DNA; or positive for hepatitis C antibody (HCVAb), Treponema pallidum antibody (TPAb/RPR), or human immunodeficiency virus antibody (HIV);
9. Pregnant or lactating patients;
10. Contraindications for MRI (e.g., metal implants such as pacemakers, claustrophobia);
11. Participation in any clinical trial involving investigational drugs within 3 months prior to dosing (or within 5 half-lives of last dose, whichever is longer);
12. Major trauma or surgery within 3 months prior to dosing, or planned surgery during the trial (excluding laparoscopy or minor procedures >4 weeks before baseline; excluding thymoma/teratoma surgery);
13. History of drug abuse or alcoholism within 1 year prior to dosing;
14. Previous treatment with stem cells or derivatives;
15. Any other condition that may increase patient risk or interfere with result interpretation, as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 38 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
DLT events | Within 24 weeks after drug administration
  Drug-related dose limiting toxicity (DLT)
mRS | 24 weeks ±10 days
  modified Ranking Scale (mRS), which ranges from 0 to 6, with higher scores indicating worse outcome, and a score of 6 representing death.

SECONDARY OUTCOMES:
AE and SAE | Within 24 weeks after drug administration
  Adverse events and severe adverse events
mRS | 5 weeks (±3 days), 12 weeks (±5 days)
  modified Ranking Scale (mRS), which ranges from 0 to 6, with higher scores indicating worse outcome, and a score of 6 representing death.
Percentage of mRS 0-2 | 5 weeks (±3 days), 12 weeks (±5 days), 24 weeks (±10 days)
  Percentage of mRS 0-2. modified Ranking Scale (mRS), which ranges from 0 to 6, with higher scores indicating worse outcome, and a score of 6 representing death.
Percentage of mRS improvement ≧ 1 | 5 weeks (±3 days), 12 weeks (±5 days), 24 weeks (±10 days)
  Percentage of mRS improvement ≧ 1. modified Ranking Scale (mRS), which ranges from 0 to 6, with higher scores indicating worse outcome, and a score of 6 representing death.
CASE score change compared to baseline | 5 weeks (±3 days), 12 weeks (±5 days), 24 weeks (±10 days)
  Clinical Assessment Scale in Autoimmune Encephalitis (CASE), ranging from 0 to 27 points, with higher score indicating more severe symptoms
ADL score change compared to baseline | 5 weeks (±3 days), 12 weeks (±5 days), 24 weeks (±10 days)
  Activity of daily living (ADL) score, ranging from 0 to 100, with higher score indicating better daily living abilities
MMSE score change compared to baseline | 5 weeks (±3 days), 12 weeks (±5 days), 24 weeks (±10 days)
  mini-mental state examination (MMSE), ranging from 0 to 30, with higher score indicating better cognition
MoCA score change compared to baseline | 5 weeks (±3 days), 12 weeks (±5 days), 24 weeks (±10 days)
  Montreal Cognitive Assessment Scale (MoCA), ranging from 0 to 30, with higher score indicating better cognition
Relapse rate of autoimmne encephalits | Within 24 weeks